CLINICAL TRIAL: NCT01893970
Title: Social Work Intervention for Adults With Mild Traumatic Brain Injury: SWIFT Pilot Study
Brief Title: SWIFT Study in the ED
Acronym: SWIFT
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Washington (Other)
Collaborators: University of California, San Francisco (Other)
Responsible Party: Principal Investigator, Megan Moore, Study Principal Investigator, University of Washington
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 44360-J
Record Dates: First submitted 2013-06-28; First posted 2013-07-09 (Estimated); Last update posted 2016-04-27 (Estimated); Status verified 2016-04

CONDITIONS: Mild Traumatic Brain Injury
MeSH Terms: conditions — Brain Concussion

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- SWIFT: Acute Social Work Intervention in the ED and Follow Up (Experimental): Participants will receive: 1) acute social work intervention for adults with mTBI, including early education, reassurance, resources and brief alcohol intervention in the ED (SWIFT-Acute) and 2) follow up telephone counseling, needs assessment and case management referral to necessary services (SWIFT).
  Interventions: Behavioral: SWIFT
- SWIFT-Acute Only: Acute social work intervention in the ED (Active Comparator): acute social work intervention for adults with mTBI, including early education, reassurance, resources and brief alcohol intervention in the ED (SWIFT-Acute)
  Interventions: Behavioral: SWIFT-Acute

INTERVENTIONS:
Behavioral: SWIFT — Participants will receive: 1) acute social work intervention for adults with mTBI, including early education, reassurance, resources and brief alcohol intervention in the ED (SWIFT-Acute) and 2) follow up telephone counseling, needs assessment and case management referral to necessary services (SWIFT).
  Arms: SWIFT: Acute Social Work Intervention in the ED and Follow Up
Behavioral: SWIFT-Acute — acute social work intervention for adults with mTBI, including early education, reassurance, resources and brief alcohol intervention in the ED (SWIFT-Acute)
  Arms: SWIFT-Acute Only: Acute social work intervention in the ED

SUMMARY:
Mild traumatic brain injury (mTBI) is a prevalent and costly public health problem with disabling consequences. More than one million civilians with mTBI are treated in US hospitals and emergency departments each year (Faul, et al., 2010). While the exact number is debated, approximately 10-15% of individuals with mTBI will experience prolonged and disabling post-concussive symptoms (Stranjalis, et al., 2008; Ruff and Weyer Jamora, 2009), and 34% will experience a psychiatric illness in the first year after injury (Fann, et al., 2004). In addition, at least 188,270 military service members sustained a TBI from 2000 to mid August 2010, and nearly 77% of these injuries were mild (Defense and Veterans Brain Injury Center, 2010). Many individuals require treatment for resulting mTBI symptoms.

The proposed study builds on preliminary research conducted by the investigators to develop and test the effectiveness of a social work delivered education and reassurance intervention for adults with mTBI (SWIFT-Acute) against usual care. The proposed study will assess acceptability and obtain preliminary effectiveness data for an enhanced social work assessment and intervention for adults with mTBI (SWIFT) discharged from the Emergency Department (ED). SWIFT includes early education, reassurance, coping strategies, resources and a brief alcohol use intervention in the ED plus follow up telephone counseling, needs assessment and case management referral to necessary services. The intervention targets cognitive, physical, psychiatric and functional outcomes; specifically, post-concussive symptoms, depression, anxiety, posttraumatic stress disorder, alcohol use, community functioning and successful linkage to community resources.

It is hypothesized that SWIFT will be acceptable to patients and that participants in the SWIFT group will report superior outcomes on measures of post-concussive symptoms, depression and anxiety, alcohol use and community functioning and will report increased successful linkages to needed resources when compared to the SWIFT-Acute group.

The specific aims of the study are:

1. Implement an innovative social work intervention for adults with mTBI (SWIFT).
2. Assess acceptability of SWIFT using qualitative interviews with participants.
3. Assess preliminary effectiveness of SWIFT compared to SWIFT-Acute alone on reduction or prevention of post-concussive symptoms, depression, anxiety, posttraumatic stress disorder (PTSD) symptoms, and alcohol use, and on improvement of community functioning and successful linkage to community resources. 80 participants will be randomized to receive SWIFT or SWIFT-Acute. Preliminary intervention effectiveness will be assessed using standard measures of post-concussive symptoms, the primary outcome, depression, anxiety, PTSD, alcohol use, and community functioning. A structured survey will be used to assess linkage to community resources.

ELIGIBILITY:
Inclusion Criteria:

Inclusion criteria are based on the World Health Organization definition of mTBI. For inclusion in the study, participants must meet following criteria:

1. At least 18 years of age and English speakers
2. Present to ED with mechanism of trauma to the head, non-penetrating injury, or recent history of trauma to the head
3. Glasgow Coma Scale score of 13-15 after 30 minutes post injury or later upon presentation for healthcare
4. Discharged from the ED in <48 hours from time of admission
5. In addition participants must have one or more of the following symptoms at time of injury:

   1. confusion or disorientation
   2. loss of consciousness for 30 minutes or less,
   3. post-traumatic amnesia for less than 24 hours
   4. other transient neurological abnormalities such as focal signs, seizure and intracranial lesion not requiring surgery

Exclusion Criteria:

1. the manifestations of mTBI are determined to be caused by penetrating craniocerebral injury
2. patients <18 years of age or non-English speaking
3. patients with intracranial lesion requiring surgery
4. patients admitted to the hospital from ED
5. patients in police custody
6. patients without a telephone contact number

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2013-04; Primary Completion 2016-07 (Estimated); Study Completion 2016-09 (Estimated)

PRIMARY OUTCOMES:
Change in Rivermead Postconcussion Symptoms Questionnaire (RPQ) | baseline, 3mo, 6mo

SECONDARY OUTCOMES:
Change in Headache Impact Test (HIT-6) | baseline, 3mo, 6mo
Change in Insomnia Severity Index (ISI) | baseline, 3mo, 6mo
Change in The Post Traumatic Stress Disorder Checklist (PCL-C) | baseline, 3mo, 6mo
Change in Cornell Service Index | baseline, 3mo, 6mo
Change in The Alcohol Use Disorders Identification Test (AUDIT) | baseline, 3mo, 6mo
Change in Community Integration Questionnaire (CIQ) | baseline, 3mo, 6mo
Change in Patient Health Questionnaire (PHQ)-9 | baseline, 3mo, 6mo
Change in Generalized Anxiety Disorder (GAD)-7 | baseline, 3mo, 6mo

OTHER OUTCOMES:
Standardized Assessment of Personality: Abbreviated Scale (SAPAS) | baseline
Change in Short Orientation Memory Concentration Test | baseline, 3mo, 6mo

CONTACTS AND LOCATIONS:
Overall Officials: Megan Moore, MSW, PHD, Principal Investigator — University of Washington
Locations (1):
- UCSF San Francisco General Hospital and Trauma Center, San Francisco, California, United States